CLINICAL TRIAL: NCT04200157
Title: Testing the Decoy Effect to Increase Tobacco Treatment Uptake
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 18-00830
Record Dates: First submitted 2019-12-13; First posted 2019-12-16 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2019-12

CONDITIONS: Tobacco Smoking
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- 1: Group assigned to the following answer combination:
  1. 2 sessions
  2. 4 sessions
  Interventions: Other: Online survey
- 2: Group assigned to the following answer combination:
  1. 2 sessions
  2. 4 sessions
  3. 7 sessions
  Interventions: Other: Online survey
- 3: Group assigned to the following answer combination:
  1. 2 sessions
  2. 7 sessions
  Interventions: Other: Online survey
- 4: Group assigned to the following answer combination:
  1. 2 sessions
  2. 7 sessions
  3. 10 sessions
  Interventions: Other: Online survey
- 5: Group assigned to the following answer combination:
  1. 2 sessions (30 minutes)
  2. 4 sessions (60 minutes)
  Interventions: Other: Online survey
- 6: Group assigned to the following answer combination:
  1. 2 sessions (30 minutes)
  2. 4 sessions (60 minutes)
  3. 7 sessions (105 minutes)
  Interventions: Other: Online survey
- 7: Group assigned to the following answer combination:
  1. 2 sessions (30 minutes)
  2. 7 sessions (105 minutes)
  Interventions: Other: Online survey
- 8: Group assigned to the following answer combination:
  1. 2 sessions (30 minutes)
  2. 7 sessions (105 minutes)
  3. 10 sessions (150 minutes)
  Interventions: Other: Online survey
- 9: Group assigned to the following answer combination:
  1. 2 sessions (30 minutes) - 10% chance of quitting
  2. 4 sessions (60 minutes) - 30% chance of quitting
  Interventions: Other: Online survey
- 10: Group assigned to the following answer combination:
  1. 2 sessions (30 minutes) - 10% chance of quitting
  2. 4 sessions (60 minutes) - 30% chance of quitting
  3. 7 sessions (105 minutes) - 30% chance of quitting
  Interventions: Other: Online survey
- 11: Group assigned to the following answer combination:
  1. 2 sessions (30 minutes) - 10% chance of quitting
  2. 7 sessions (105 minutes) - 30% chance of quitting
  Interventions: Other: Online survey
- 12: Group assigned to the following answer combination:
  1. 2 sessions (30 minutes) - 10% chance of quitting
  2. 7 sessions (105 minutes) - 30% chance of quitting
  3. 10 sessions (150 minutes) - 30% chance of quitting
  Interventions: Other: Online survey

INTERVENTIONS:
Other: Online survey — Subjects will complete a single survey that takes 5-10 minutes to complete

SUMMARY:
Prior research has shown that the context in which program options are presented to consumer impacts consumer choice (known as the 'decoy effect'). The aims of this study are to: (1) test whether the decoy effect can impact smokers' selection of hypothetical tobacco treatment options; (2) examine sociodemographic moderators of the decoy effect; and and (3) examine whether presenting the time and clinical effectiveness of of the different treatment options modifies the decoy effect.

DETAILED DESCRIPTION:
The investigators will recruit and conduct a cross-sectional online survey through ResearchMatch (www.researchmatch.org) with 600 tobacco users across the country. The survey will ask participants for their preferences regarding hypothetical tobacco treatment programs. Participants will be randomized to 12 conditions (n=50 per condition). Each condition has a different combination of treatment options. The survey will also assess sociodemographics and tobacco use behaviors. All participants will be asked if they would like to receive information about the state's smoking cessation quitline. Participants who would like to receive information will be given the 1800-QUIT-NOW number and smokefree.gov website address.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported current tobacco use

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from ResearchMatch.org. People who are in ResearchMatch.org's database will be eligible if they are 18 years or older and self-report current tobacco use.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Number of counseling calls chosen | 6 months
Number of weeks until quit date chosen | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Langone Health - Translational Research Building, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rogers ES, Vargas EA, Voigt E. Exploring the decoy effect to guide tobacco treatment choice: a randomized experiment. BMC Res Notes. 2020 Jan 2;13(1):3. doi: 10.1186/s13104-019-4873-0. PMID 31898550